CLINICAL TRIAL: NCT03018405
Title: A Multi-national, Open-label, Dose Escalation Phase I Study to Assess the Safety and Clinical Activity of Multiple Administrations of NKR-2 in Patients With Different Metastatic Tumor Types (THINK - THerapeutic Immunotherapy With NKR-2)
Brief Title: A Dose Escalation Phase I Study to Assess the Safety and Clinical Activity of Multiple Cancer Indications
Acronym: THINK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2T-002
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2018-11

CONDITIONS: Acute Myeloid Leukemia/Myelodysplastic Syndrome; Multiple Myeloma (MM)
MeSH Terms: conditions — GATA2 Deficiency; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: The maximum number of patients to be enrolled is 146:
  * 36 in the dose escalation segment (cohorts 1-6, 18 per arm),
  * 24 in the additional cohorts 8-11 (12 per arm),
  * 86 patients in the Phase I expansion segment (note that the analysis of this segment will also include a maximum of 12 additional patients from the dose escalation segment).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hematological tumors (Experimental): The dose escalation arm for hematological tumors will use a 3 +3 design to determine the maximum tolerated dose. Two additional cohorts will be added in this dose escalation arm with the aim to provide a more intense treatment during the induction treatment (cycle 1 of injection). Cohort 10-11 (only in AML/MDS) will evaluate a tighter schedule of NKR-2 injections at 1x109 or potentially 3x109 NKR-2 per injection with the three first injections within the induction cycle (cycle 1) separated by a 1-week interval followed two weeks later by a second cycle (cycle 2) with a 2-weeks interval between each three NKR 2 injections.
  Interventions: Biological: NKR-2 cells
- Solid Tumors (Experimental): The dose escalation arm for solid tumors will use a 3 +3 design to determine the maximum tolerated dose. Two additional cohorts will be added in this dose escalation arm with the aim to provide a more intense treatment during the induction treatment (cycle 1 of injection). Cohort cohort 8-9 ( only in CRC) will evaluate a tighter schedule of NKR-2 injections at 1x109 or potentially 3x109 NKR-2 per injection with the three first injections within the induction cycle (cycle 1) separated by a 1-week interval followed two weeks later by a second cycle (cycle 2) with a 2-weeks interval between each three NKR 2 injections.
  Interventions: Biological: NKR-2 cells

INTERVENTIONS:
Biological: NKR-2 cells — In cohorts 1-6, the schedule of administration will be 3 NKR-2 doses administered with a 2-week interval. In absence of progressive disease at the first tumor assessment following NKR-2 administration (on Visit D29 for hematological tumors or on Visit D57 for solid tumors), and according to product availability, the patient will receive a new cycle of 3 administrations maximum with a 2-week interval, at a dose of 1x109 NKR-2 cells per injection, or at the same dose of cycle 1 if it was below 1x109 NKR-2 cells.
  Patients in cohorts 8-9 (solid arm) and 10-11 (hematological arm) of first segment will receive 3 treatment doses at 1x109 NKR-2 (cohorts 8 and 10) or 3x109 NKR-2 (cohorts 9 and 11) per injection, with a 1-week interval between each dose. A second cycle of three NKR-2 injections at the same dose as in 1st cycle will be administered 2 weeks after the third NKR-2 injection, and with a 2-week interval between each dose.
  Other Names: NKG2D-CAR construct

SUMMARY:
THINK (THerapeutic Immunotherapy with NKR-2) is a multinational (EU/US) open-label Phase I study to assess the safety and clinical activity of multiple administrations of autologous NKR-2 cells in seven refractory cancers, including five solid tumors (colorectal, ovarian, bladder, triple-negative breast and pancreatic cancers) and two hematological tumors (acute myeloid leukemia and multiple myeloma).

DETAILED DESCRIPTION:
This open-label Phase I study aims at assessing the safety and clinical activity of the NKR-2 treatment administered 3 times with a 2-week interval between each administration in different tumor types. In absence of progressive disease at the first tumor assessment following NKR-2 administratio, the patient will receive a new cycle of 3 administrations maximum with a 2-week interval. The study will contain two consecutive segments: a Phase I dose escalation and a Phase I expansion segment.

The Phase I dose escalation segment will include 2 arms, one in solid tumors and one in hematological tumors. The dose escalation design will include 3 dose levels: The dose escalation phase will consist of 3 cohorts (Cohorts 1-3) for the solid tumors, and 3 cohorts (Cohorts 4-6) for the hematological tumors; with each set of 3 cohorts receiving escalating doses of the NKR-2 therapy.

Two additional cohorts will be added in each dose escalation arm with the aim to provide a more intense treatment during the induction treatment. These additional cohorts in both the solid arm (cohort 8-9 - only in CRC) and in the hematological arm of the study (cohort 10-11 - only in AML/MDS) will therefore evaluate a tighter schedule of NKR-2 injections with the three first injections within the induction cycle separated by a 1-week interval followed two weeks later by a second cycle (cycle 2) with a 2-weeks interval between each three NKR 2 injections. These cohorts will each enroll 3 patients in case of no DLT. Based on safety and early clinical data from these cohorts, the specific schedule of cohorts 8-11 might be selected for the expansion.

ELIGIBILITY:
Main inclusion criteria are:

* Men or women ≥ 18 years old at the time of signing the ICF,
* Patient with a CRC, epithelial ovarian cell or fallopian tube carcinoma, urothelial carcinoma, TNBC, pancreatic cancer, AML/MDS or MM,
* Disease must be measurable according to the corresponding guidelines,
* Patient with an ECOG performance status 0 or 1, and AML patients with anemia resulting in an ECOG performance status of 2,
* Patient with adequate bone marrow reserve, hepatic and renal functions.
* Patients must have sufficient pulmonary functions with a Forced Expiratory Volume in the first second (FEV-1)/Forced Vital Capacity (FVC) ≥ 0.7 with FEV-1 ≥ 50% predicted.

Main exclusion criteria are:

* Patient with a tumor metastasis in the central nervous system,
* Patients who have received another cancer therapy within 2 weeks before the planned day for the apheresis (except hydroxyurea for AML patients),
* Patients who receive or are planned to receive any other investigational product within the 3 weeks before the planned day for the first NKR-2 administration (except hydroxyurea for AML patients),
* Patient is under systemic immunosuppressive drugs, unless specific cases authorized per protocol,
* Patients who have received other cell therapies,
* Patients who underwent major surgery within 4 weeks before the planned day for the first NKR-2 administration.
* Patient cannot present with history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis and/or active or acute exacerbation of chronic obstructive pulmonary disease (COPD).

Detailed disease specific criteria exist and can be discussed with contacts listed below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of NKR-2 infusion | 24 months
  Safety defined by Occurrence of adverse events (AEs) and serious adverse events (SAEs) during the study treatment until 30 days after the last study treatment administration.

SECONDARY OUTCOMES:
Clinical activity of the treatment in each tumor type | 24 months
  Clinical activity of the treatment in each tumor type

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lehmann, MD, Principal Investigator — Celyad Oncology SA
Locations (4):
- United States (2):
  - Tampa, Florida
  - Buffalo, New York
- Belgium (2):
  - Brussels
  - Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sallman DA, Kerre T, Havelange V, Poire X, Lewalle P, Wang ES, Brayer JB, Davila ML, Moors I, Machiels JP, Awada A, Alcantar-Orozco EM, Borissova R, Braun N, Dheur MS, Gilham DE, Lonez C, Lehmann FF, Flament A. CYAD-01, an autologous NKG2D-based CAR T-cell therapy, in relapsed or refractory acute myeloid leukaemia and myelodysplastic syndromes or multiple myeloma (THINK): haematological cohorts of the dose escalation segment of a phase 1 trial. Lancet Haematol. 2023 Mar;10(3):e191-e202. doi: 10.1016/S2352-3026(22)00378-7. Epub 2023 Feb 7. PMID 36764323
- [Derived] Lonez C, Verma B, Hendlisz A, Aftimos P, Awada A, Van Den Neste E, Catala G, Machiels JH, Piette F, Brayer JB, Sallman DA, Kerre T, Odunsi K, Davila ML, Gilham DE, Lehmann FF. Study protocol for THINK: a multinational open-label phase I study to assess the safety and clinical activity of multiple administrations of NKR-2 in patients with different metastatic tumour types. BMJ Open. 2017 Nov 12;7(11):e017075. doi: 10.1136/bmjopen-2017-017075. PMID 29133316